CLINICAL TRIAL: NCT06560164
Title: Restrictive Versus Liberal Thresholds for Red Blood Cell Transfusion in ExtraCorporeal Membrane Oxygenation - the TREC Study
Brief Title: Restrictive Versus Liberal Thresholds for RBC Transfusion in ECMO
Acronym: TREC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, A.P.J. Vlaar, Prof. Dr., Amsterdam UMC, location AMC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL84295.018.23; NL84295.018.23 (Other: IRB Amsterdam UMC); 84295 (Other: ABR (Dutch: General Assessment and Registration Form)); B3222022001258 (Registry Identifier: Belgium Registration Number); 2023-07691-01 (Registry Identifier: Swedish Registration Number); 10390032310031 (Other Grant/Funding Number: ZonMW)
Record Dates: First submitted 2024-08-13; First posted 2024-08-19 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Transfusion; Red Blood Cell; Extracorporeal Membrane Oxygenation; Anemia; ECMO
Keywords: Transfusion; Red Blood Cell; Extracorporeal Membrane Oxygenation; Anemia; ECMO
MeSH Terms: conditions — Anemia | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Intervention Model Description: Study design: This is a non-inferiority, randomized controlled trial in patients receiving ECMO.
  Study population: Patients, 18 years or older, receiving ECMO (see additional details below).
  Randomization will be stratified by:
  * Center;
  * ECMO mode, divided by:
    * VV ECMO (or triple cannulation methods with primarily a pulmonary indication);
    * VA ECMO (or triple cannulation methods with primarily a cardiac indication or extracorporeal cardiopulmonary resuscitation [ECPR]).
  Intervention:
  1. Restrictive RBC transfusion threshold: in case the Hb transfusion trigger of 7.0 g/dL (4.3 mmol/L) is reached, 1 RBC unit at a time will be transfused.
  2. Liberal RBC transfusion threshold: in case the Hb transfusion trigger of 9.0 g/dL (5.6 mmol/L) is reached, 1 RBC unit at a time will be transfused.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Restrictive strategy (Active Comparator): The restrictive strategy will consist of a transfusion Hb threshold of 7.0 g/dL, with a target Hb range of 7.1 - 9.0 g/dL. These thresholds are based on previous non-inferior trials in the patient populations in which VV ECMO (comparable to sepsis) and VA ECMO (cardiac surgery, acute myocardial infarction) are often applied.
  Interventions: Other: Red Blood Cell transfusion
- Liberal strategy (Active Comparator): The liberal strategy will consist of a transfusion Hb threshold of 9.0 g/dL, with a target Hb range of 9.1 - 11.0 g/dL. These Hb thresholds are based on thresholds that are currently used in ECMO.
  Interventions: Other: Red Blood Cell transfusion

INTERVENTIONS:
Other: Red Blood Cell transfusion — When the appropriate Hb threshold is reached, patients in each group will have one unit of RBC administered at a time. Within 3 hours after the transfusion, a repeat Hb concentration will be measured. Each group will only be transfused when their Hb level falls below the transfusion threshold. In case of a outlier measurement, clinicians are advised to repeat the measurement. The RBC transfusion must take place within 4 hours when the Hb trigger was measured.
  Other Names: RBC transfusion; pRBCs; packed Red Blood Cells

SUMMARY:
Rationale: In patients supported with extracorporeal membrane oxygenation (ECMO), transfusion of red blood cells (RBC) is very common. This is possibly due to the application of liberal thresholds and the lack of evidence-based guidelines. Although RBC transfusion can be lifesaving, it is also a risk-bearing intervention with substantial risk for morbidity and mortality in this critically ill population. Also, with increasing scarcity, RBC transfusions are becoming more expensive. Furthermore, in the past decades it has been shown in several critically ill patient populations - not on ECMO - that maintaining a restrictive hemoglobin (Hb) threshold for RBC transfusion is non-inferior, including in cardiothoracic surgery, acute myocardial infarction and septic shock. Therefore, the investigators hypothesize that a restrictive transfusion threshold for RBC is safe to apply in patients on ECMO in comparison with a liberal transfusion threshold.

Objective: The primary objective of this trial is to study in a prospective randomized comparison whether a restrictive RBC transfusions strategy is non-inferior compared to a liberal strategy in patients on ECMO with respect to 90-day mortality.

Study design: Prospective multi-center randomized controlled non-inferiority trial.

Study population: Patients, 18 years or older, receiving ECMO.

Intervention: Restrictive RBC transfusion threshold: in case the Hb transfusion trigger of 7.0 g/dL (4.3 mmol/L) is reached, 1 RBC unit at a time will be transfused. The aimed Hb target range of the restrictive/intervention group will be 7.1 - 9.0 g/dL (4.3 - 5.6 mmol/L). Liberal RBC transfusion threshold: in case the Hb transfusion trigger of 9.0 g/dL (5.6 mmol/L) is reached, 1 RBC unit at a time will be transfused. Target range of the liberal group is defined as Hb 9.1 - 11.0 g/dL

Main study parameters/endpoints: The primary outcome parameter is 90-day all-cause mortality.

Secondary outcomes include: 1) proportion of patients on ECMO exposed to allogeneic RBC transfusion; 2) RBC volume infused per patient during ECMO; 3) reasons for RBC transfusion other than Hb triggers; 4) transfusion reactions; 5) time on ECMO; 6) length of hospital- and ICU-stay; 7) in-ICU morbidity; 8) quality of life (QoL), iMTA Medical Consumption Questionnaire (iMCQ) and Productivity Cost Questionnaire (iPCQ) at 3, 6, 9, and 12 months; 9) costs related to a) transfusion, b) hospital admission and c) transfusion-related sequelae.

DETAILED DESCRIPTION:
Extracorporeal membrane oxygenation (ECMO) is used as a supportive method in case of temporary and potentially reversible cardiac or respiratory failure, refractory to conventional therapies. Over the past decades, application of ECMO has been increasing worldwide. As ECMO is generally used as a 'last resort' therapy, the population is vulnerable, and many complications can occur. Anemia occurs in >90% of the patients on ECMO, caused by many different patient-related, disease-related, and ECMO-related factors. Nevertheless, rationale for the recommended hemoglobin (Hb) thresholds for red blood cell (RBC) transfusion in this patient population is limited. This was recently confirmed by the members of the European Society of Intensive Care Medicine (ESICM), who concluded in their clinical practice guideline that no recommendation on transfusion thresholds can be made, since solid evidence is missing. The panel stated that this area is a research priority.

This lack of evidence-based guidelines may explain the high variance in Hb thresholds applied, as well as the thresholds in use being relatively liberal. As a result, transfusion of RBC is very common. Observational studies describe that almost 9 out of 10 patients receiving ECMO receive at least one RBC transfusion, and the total amount is very high. These numbers are even more remarkable when comparing to other patient populations in the Intensive Care Unit (ICU), in which 1 out of 4 patients receives RBC with way lesser amounts. One of the main arguments for using a liberal transfusion threshold in ECMO is the hypothesis that in patients receiving ECMO, tissue hypoxemia can develop due to decreased pulmonary oxygen intake (e.g., in pneumonia as indication for veno-venous [VV] ECMO), or decreased cardiac output (e.g., in myocardial infarction as indication for veno-arterial [VA] ECMO). By providing a larger Hb buffer, it is assumed that the oxygen delivery (DO2) will be preserved and the incidence of tissue hypoxemia will be reduced. However, evidence to either confirm or refute this hypothesis is lacking. Since ECMO ensures oxygenation and can provide a blood flow of up to 7 L/min, it can be assumed that ECMO fully compensates for the possible decrease in DO2.

Although RBC transfusion can be lifesaving, it is also a risk-bearing intervention with substantial risk for morbidity and mortality in this critically ill population. In similar patient populations without ECMO, maintaining a restrictive RBC transfusion strategy (Hb 7.0 g/dL) has been proven non-inferior to a more liberal practice (Hb 9.0 g/dL). This includes randomized controlled trials (RCTs) in septic shock patients (comparable to patients on VV ECMO), cardiothoracic surgery patients, and even patients suffering from acute myocardial infarction and anemia (comparable to patients on VA ECMO). Although these conclusions are promising, they cannot directly be translated to patients supported by ECMO, although underlying conditions are similar. Moreover, RBC transfusions are expensive and donors are becoming more scarce. In this vulnerable critically ill patient population with an enhanced risk for transfusion related complications, it is of utmost importance to only administer a RBC transfusion when the benefits outweigh the risks.

As both anemia and transfusion are associated with poor outcomes, observational studies cannot answer the question whether a restrictive Hb threshold is non-inferior to a liberal strategy. There is a need to define general thresholds to improve the efficiency of indications for RBC transfusion in ECMO. Since one of the most commonly used triggers for RBC transfusion is Hb concentration, this forms the basis for our study to investigate whether it is non-inferior to maintain a restrictive transfusion threshold (intervention group: Hb 7 g/dL) compared to the current standard of 9 g/dL in patients on ECMO, independent of the mode.

This study is funded by ZonMW (Zorgonderzoek Medische Wetenschappen), part of the NWO (Nederlandse Organisatie voor Wetenschappelijk Onderzoek; the Dutch Organization for Scientific Research, Den Haag, the Netherlands), reference number 10390032310031.

ELIGIBILITY:
Inclusion Criteria:

* Patient is aged 18 years or older;
* Is receiving ECMO;
* (Deferred) informed consent.

Exclusion Criteria:

* Not expected to survive for 24 hours when assessed;
* Inability to receive blood products;
* (Known) decline to blood transfusions (e.g., Jehovah's Witnesses);
* Extracorporeal carbon dioxide removal (ECCO2R) using low blood flow devices or pumpless devices (i.e., MINILUNG ®, PrismaLung+);
* Received ECMO over 48h before screening for eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
90-day all-cause mortality | 90 days
  The primary outcome measure is all-cause mortality within 90 days, i.e. the proportion of patients who die from any cause during this 90-day period following ECMO support.

SECONDARY OUTCOMES:
In-hospital mortality | 30 days
  All-cause mortality during the hospital stay refers to the proportion of patients who died from any cause while they were still admitted to the hospital.
Duration | 30 days
  The duration of ECMO support, along with the length of ICU and hospital stays, are key metrics that quantify the total time a patient receives ECMO treatment, is in the intensive care unit, and remains in the hospital, measured in both days and hours.
Red blood cell transfusion exposure | 30 days
  The proportion of patients on ECMO who receive allogeneic red blood cell (RBC) transfusions.
Adherence | 30 days
  The number of adherence and non-adherence transfusion events.
EQ-5D-5L | 3, 6, 9, and 12 months
  A quality of life questionnaire assessing various domains including mobility, self-care, daily activities, and pain/discomfort, as well as emotional states like fear/sadness. Each domain is rated on a 5-point scale, where 1 indicates no problems and 5 indicates severe problems. Additionally, the questionnaire includes a EuroQol Visual Analogue Scale (EQ-VAS), which is a vertical scale ranging from 100 (best imaginable health) to 0 (worst imaginable health).
Medical Consumption | 3, 6, 9, and 12 months
  The iMTA Medical Consumption Questionnaire (iMCQ) will be used to assess medical consumption and associated costs during the first year following ECMO support. This questionnaire collects detailed information on healthcare utilization, such as hospital visits, medications, medical procedures, and other related services, enabling an analysis of the overall costs incurred during the recovery period. The iMCQ does not include an outcome scale but focuses solely on quantifying the extent and cost of medical resources used.
Productivity Cost | 3, 6, 9, and 12 months
  The Productivity Cost Questionnaire (iPCQ) will be utilized to assess productivity loss during the first year following ECMO support. This questionnaire captures data on absenteeism, reduced efficiency at work, and lost productivity due to health-related issues. The iPCQ focuses exclusively on quantifying the extent of productivity loss without including an outcome scale, providing a clear picture of the economic impact associated with recovery in the first year post-ECMO.

OTHER OUTCOMES:
In-ICU morbidity | 30 days
  All in-ICU morbidity, including neurological, cardiac, hemorrhagic, abdominal, renal, infection, peripheral, and transfusion-related complications.
Transfusion reasons | 30 days
  To evaluate the reasons for RBC transfusion beyond solely using hemoglobin (Hb) levels as the trigger.
Exposure to other transfusion products | 30 days
  The number of transfusions of other blood-derived products or coagulation factors, such as platelet concentrates.
Supportive therapy duration | 30 days
  The duration of supportive therapies, including invasive mechanical ventilation and renal replacement therapy, measured in both days and hours.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander P.J. Vlaar, PhD, Principal Investigator — Amsterdam UMC, location AMC
Locations (12):
- Belgium (4):
  - Hôpital Erasme Brussels, Brussels, Brussels Capital
  - KU Leuven, medical IC, Leuven, Flemish Brabant
  - KU Leuven, surgical IC, Leuven, Flemish Brabant
  - CHU Charleroi, Charleroi, Hainaut
- Netherlands (7):
  - Medisch Spectrum Twente (MST), Enschede, Drenthe
  - Maastricht Universitair Medisch Centrum+ (MUMC+), Maastricht, Limburg
  - Amsterdam UMC, location AMC, Amsterdam, North Holland
  - Universitair Medisch Centrum Groningen (UMCG), Groningen, Provincie Groningen
  - Leids Universitair Medisch Centrum (LUMC), Leiden, South Holland
  - Erasmus MC, Rotterdam, South Holland
  - St. Antonius Ziekenhuis, Nieuwegein, Utrecht
- Karolinska Universtiy Hospital, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be submitted for publication in a prominent journal.
Supporting Information: Study Protocol
Time Frame: The protocol will be available after publication, expected within 1 year after the start of all participating centers.
Access Criteria: Open access.
URL: https://ecmo-nl.com/trec.html

REFERENCES:
- [Background] Gattinoni L, Carlesso E, Langer T. Clinical review: Extracorporeal membrane oxygenation. Crit Care. 2011;15(6):243. doi: 10.1186/cc10490. Epub 2011 Dec 8. PMID 22188792
- [Background] Makdisi G, Wang IW. Extra Corporeal Membrane Oxygenation (ECMO) review of a lifesaving technology. J Thorac Dis. 2015 Jul;7(7):E166-76. doi: 10.3978/j.issn.2072-1439.2015.07.17. PMID 26380745
- [Background] Vlaar AP, Oczkowski S, de Bruin S, Wijnberge M, Antonelli M, Aubron C, Aries P, Duranteau J, Juffermans NP, Meier J, Murphy GJ, Abbasciano R, Muller M, Shah A, Perner A, Rygaard S, Walsh TS, Guyatt G, Dionne JC, Cecconi M. Transfusion strategies in non-bleeding critically ill adults: a clinical practice guideline from the European Society of Intensive Care Medicine. Intensive Care Med. 2020 Apr;46(4):673-696. doi: 10.1007/s00134-019-05884-8. Epub 2020 Jan 7. PMID 31912207
- [Background] de Bruin S, Scheeren TWL, Bakker J, van Bruggen R, Vlaar APJ; Cardiovascular Dynamics Section and Transfusion Guideline Task Force of the ESICM. Transfusion practice in the non-bleeding critically ill: an international online survey-the TRACE survey. Crit Care. 2019 Sep 11;23(1):309. doi: 10.1186/s13054-019-2591-6. PMID 31511083
- [Background] Martucci G, Grasselli G, Tanaka K, Tuzzolino F, Panarello G, Schmidt M, Bellani G, Arcadipane A. Hemoglobin trigger and approach to red blood cell transfusions during veno-venous extracorporeal membrane oxygenation: the international TRAIN-ECMO survey. Perfusion. 2019 Apr;34(1_suppl):39-48. doi: 10.1177/0267659119830526. PMID 30966906
- [Background] Aubron C, DePuydt J, Belon F, Bailey M, Schmidt M, Sheldrake J, Murphy D, Scheinkestel C, Cooper DJ, Capellier G, Pellegrino V, Pilcher D, McQuilten Z. Predictive factors of bleeding events in adults undergoing extracorporeal membrane oxygenation. Ann Intensive Care. 2016 Dec;6(1):97. doi: 10.1186/s13613-016-0196-7. Epub 2016 Oct 6. PMID 27714705
- [Background] Raasveld SJ, Karami M, van den Bergh WM, Oude Lansink-Hartgring A, van der Velde F, Maas JJ, van de Berg P, de Haan M, Lorusso R, Delnoij TSR, Dos Reis Miranda D, Mandigers L, Scholten E, Overmars M, Silvio Taccone F, Brasseur A, Dauwe DF, De Troy E, Hermans G, Meersseman P, Pappalardo F, Fominskiy E, Ivancan V, Bojcic R, de Metz J, van den Bogaard B, Donker DW, Meuwese CL, de Bakker M, Reddi B, de Bruin S, Lagrand WK, Henriques JPS, Broman LM, Vlaar APJ. RBC Transfusion in Venovenous Extracorporeal Membrane Oxygenation: A Multicenter Cohort Study. Crit Care Med. 2022 Feb 1;50(2):224-234. doi: 10.1097/CCM.0000000000005398. PMID 35100195
- [Background] Vincent JL, Baron JF, Reinhart K, Gattinoni L, Thijs L, Webb A, Meier-Hellmann A, Nollet G, Peres-Bota D; ABC (Anemia and Blood Transfusion in Critical Care) Investigators. Anemia and blood transfusion in critically ill patients. JAMA. 2002 Sep 25;288(12):1499-507. doi: 10.1001/jama.288.12.1499. PMID 12243637
- [Background] Bosboom JJ, Klanderman RB, Zijp M, Hollmann MW, Veelo DP, Binnekade JM, Geerts BF, Vlaar APJ. Incidence, risk factors, and outcome of transfusion-associated circulatory overload in a mixed intensive care unit population: a nested case-control study. Transfusion. 2018 Feb;58(2):498-506. doi: 10.1111/trf.14432. Epub 2017 Dec 13. PMID 29238981
- [Background] Hebert PC, Wells G, Blajchman MA, Marshall J, Martin C, Pagliarello G, Tweeddale M, Schweitzer I, Yetisir E. A multicenter, randomized, controlled clinical trial of transfusion requirements in critical care. Transfusion Requirements in Critical Care Investigators, Canadian Critical Care Trials Group. N Engl J Med. 1999 Feb 11;340(6):409-17. doi: 10.1056/NEJM199902113400601. PMID 9971864
- [Background] Mazer CD, Whitlock RP, Fergusson DA, Hall J, Belley-Cote E, Connolly K, Khanykin B, Gregory AJ, de Medicis E, McGuinness S, Royse A, Carrier FM, Young PJ, Villar JC, Grocott HP, Seeberger MD, Fremes S, Lellouche F, Syed S, Byrne K, Bagshaw SM, Hwang NC, Mehta C, Painter TW, Royse C, Verma S, Hare GMT, Cohen A, Thorpe KE, Juni P, Shehata N; TRICS Investigators and Perioperative Anesthesia Clinical Trials Group. Restrictive or Liberal Red-Cell Transfusion for Cardiac Surgery. N Engl J Med. 2017 Nov 30;377(22):2133-2144. doi: 10.1056/NEJMoa1711818. Epub 2017 Nov 12. PMID 29130845
- [Background] Murphy GJ, Pike K, Rogers CA, Wordsworth S, Stokes EA, Angelini GD, Reeves BC; TITRe2 Investigators. Liberal or restrictive transfusion after cardiac surgery. N Engl J Med. 2015 Mar 12;372(11):997-1008. doi: 10.1056/NEJMoa1403612. PMID 25760354
- [Background] Ducrocq G, Gonzalez-Juanatey JR, Puymirat E, Lemesle G, Cachanado M, Durand-Zaleski I, Arnaiz JA, Martinez-Selles M, Silvain J, Ariza-Sole A, Ferrari E, Calvo G, Danchin N, Avendano-Sola C, Frenkiel J, Rousseau A, Vicaut E, Simon T, Steg PG; REALITY Investigators. Effect of a Restrictive vs Liberal Blood Transfusion Strategy on Major Cardiovascular Events Among Patients With Acute Myocardial Infarction and Anemia: The REALITY Randomized Clinical Trial. JAMA. 2021 Feb 9;325(6):552-560. doi: 10.1001/jama.2021.0135. PMID 33560322
- [Background] Kracalik I, Mowla S, Basavaraju SV, Sapiano MRP. Transfusion-related adverse reactions: Data from the National Healthcare Safety Network Hemovigilance Module - United States, 2013-2018. Transfusion. 2021 May;61(5):1424-1434. doi: 10.1111/trf.16362. Epub 2021 Apr 20. PMID 33880771
- [Background] Holst LB, Haase N, Wetterslev J, Wernerman J, Aneman A, Guttormsen AB, Johansson PI, Karlsson S, Klemenzson G, Winding R, Nebrich L, Albeck C, Vang ML, Bulow HH, Elkjaer JM, Nielsen JS, Kirkegaard P, Nibro H, Lindhardt A, Strange D, Thormar K, Poulsen LM, Berezowicz P, Badstolokken PM, Strand K, Cronhjort M, Haunstrup E, Rian O, Oldner A, Bendtsen A, Iversen S, Langva JA, Johansen RB, Nielsen N, Pettila V, Reinikainen M, Keld D, Leivdal S, Breider JM, Tjader I, Reiter N, Gottrup U, White J, Wiis J, Andersen LH, Steensen M, Perner A. Transfusion requirements in septic shock (TRISS) trial - comparing the effects and safety of liberal versus restrictive red blood cell transfusion in septic shock patients in the ICU: protocol for a randomised controlled trial. Trials. 2013 May 23;14:150. doi: 10.1186/1745-6215-14-150. PMID 23702006
- [Background] Hayden SJ, Albert TJ, Watkins TR, Swenson ER. Anemia in critical illness: insights into etiology, consequences, and management. Am J Respir Crit Care Med. 2012 May 15;185(10):1049-57. doi: 10.1164/rccm.201110-1915CI. Epub 2012 Jan 26. PMID 22281832
- [Background] Carson JL, Stanworth SJ, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding allogeneic red blood cell transfusion. Cochrane Database Syst Rev. 2016 Oct 12;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub4. PMID 27731885
- [Background] Docherty AB, Turgeon AF, Walsh TS. Best practice in critical care: anaemia in acute and critical illness. Transfus Med. 2018 Apr;28(2):181-189. doi: 10.1111/tme.12505. Epub 2018 Jan 25. PMID 29369437
- [Background] Spinelli E, Bartlett RH. Anemia and Transfusion in Critical Care: Physiology and Management. J Intensive Care Med. 2016 Jun;31(5):295-306. doi: 10.1177/0885066615571901. Epub 2015 Feb 18. PMID 25693602
- [Background] Gong MN, Thompson BT, Williams P, Pothier L, Boyce PD, Christiani DC. Clinical predictors of and mortality in acute respiratory distress syndrome: potential role of red cell transfusion. Crit Care Med. 2005 Jun;33(6):1191-8. doi: 10.1097/01.ccm.0000165566.82925.14. PMID 15942330
- [Background] Corwin HL, Gettinger A, Pearl RG, Fink MP, Levy MM, Abraham E, MacIntyre NR, Shabot MM, Duh MS, Shapiro MJ. The CRIT Study: Anemia and blood transfusion in the critically ill--current clinical practice in the United States. Crit Care Med. 2004 Jan;32(1):39-52. doi: 10.1097/01.CCM.0000104112.34142.79. PMID 14707558
- [Background] Vlaar APJ, Toy P, Fung M, Looney MR, Juffermans NP, Bux J, Bolton-Maggs P, Peters AL, Silliman CC, Kor DJ, Kleinman S. A consensus redefinition of transfusion-related acute lung injury. Transfusion. 2019 Jul;59(7):2465-2476. doi: 10.1111/trf.15311. Epub 2019 Apr 16. PMID 30993745
- [Background] Wiersum-Osselton JC, Whitaker B, Grey S, Land K, Perez G, Rajbhandary S, Andrzejewski C Jr, Bolton-Maggs P, Lucero H, Renaudier P, Robillard P, Santos M, Schipperus M. Revised international surveillance case definition of transfusion-associated circulatory overload: a classification agreement validation study. Lancet Haematol. 2019 Jul;6(7):e350-e358. doi: 10.1016/S2352-3026(19)30080-8. Epub 2019 May 9. PMID 31080132
- See also: Extracorporeal Life Support Organization. Extracorporeal Life Support Organization ECLS Registry Report Overall Outcomes. 2019 — https://www.elso.org/Registry/Statistics/InternationalSummary.aspx
- See also: Additional study information and progress overview — https://ecmo-nl.com/trec.html